CLINICAL TRIAL: NCT05511623
Title: Efficacy and Safety of Tislelizumab Combined With Concurrent Chemoradiotherapy as First-line Treatment for Stage IIIC2 Cervical Cancer
Brief Title: Tislelizumab Combined With Concurrent Chemoradiotherapy as First-line Treatment for Stage IIIC2 Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W2022
Record Dates: First submitted 2022-07-13; First posted 2022-08-23 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
Keywords: cervical carcinoma; PD-1; chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tislelizumab; spartalizumab; Chemoradiotherapy; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized (1:1) to Arm A or Arm B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tislelizumab (Experimental): The external radiation is administered at 45-50Gy/25f and brachytherapy is performed sequentially at 6Gy/time to a total doses of 30 Gy. The concomitant chemotherapy regimen is cisplatin 40mg/m2 on day 1 once every week for 5 weeks. In addition, patients also receive tislelizumab (200 mg, day 1) once every 3 weeks until disease progression or intolerable toxicity occurs or one year.
  Interventions: Drug: tislelizumab
- concurrent chemoradiotherapy (Active Comparator): The external radiation is administered at 45-50Gy/25f and brachytherapy is performed sequentially at 6Gy/time to a total doses of 30 Gy. The concomitant chemotherapy regimen is cisplatin 40mg/m2 on day 1 once every week for 5 weeks.
  Interventions: Other: concurrent chemoradiotherapy

INTERVENTIONS:
Drug: tislelizumab — standard radiotherapy with concomitant cisplatin 40mg/m2 once every week for 5 weeks, combined with tislelizumab (200 mg, day 1) once every 3 weeks until disease progression or intolerable toxicity occurs or one year.
  Other Names: pd-1 antibody
  Arms: tislelizumab
Other: concurrent chemoradiotherapy — standard radiotherapy with concomitant cisplatin 40mg/m2 on day 1 once every week for 5 weeks.
  Other Names: DDP combined with radiotherapy
  Arms: concurrent chemoradiotherapy

SUMMARY:
To evaluate the efficacy and safety of tislelizumab combined with concurrent chemoradiotherapy in first-line treatment of stage IIIC2 cervical cancer.

DETAILED DESCRIPTION:
This is a multicenter, prospective, and randomized phase II clinical trial. Patients assigned to experimental group will receive standard radiotherapy with concomitant cisplatin 40mg/m2 once every week for 5 weeks, combined with tislelizumab (200 mg, day 1) once every 3 weeks until disease progression or intolerable toxicity occurs or one year. Patients assigned to control group will undergo standard radiotherapy with concomitant cisplatin 40mg/m2 once every week for 5 weeks. Compare the efficacy and toxicity of the two regimens in patients with stage IIIC2 cervical cancer.

ELIGIBILITY:
Inclusion criteria:

(1)18-70 years old; (2)Histologically confirmed squamous carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix; (3)Patients with 2018 FIGO stage IIIC2 cervical cancer; (4)At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1; (5)Eastern Cooperative Oncology Group score 0-1; (6)No metastatic diseases; (7)Must have an average life expectancy of 6 months; (8)Participants must have normal organ and marrow function as defined below: (hemoglobin ≥90g/L,neutrophils ≥1.5×109/L, platelets ≥80×109/L, ALB≥30g/L, Total bilirubin≤1.5 x institutional upper limit of normal, AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal, Creatinine clearance≥60 mL/min; (9)Patients with menopause, or patients of reproductive potential were required to take effective contraceptive measures for the duration of the study and had a negative pregnancy test result, non-lactating women; (10)Patients volunteered to participate in the study and sign the informed consent.

Exclusion criteria:

1. Diagnosed with any other cancer within the past 5 years;
2. Known allergy to any component of the drug;
3. Congenital or acquired immune deficiency (such as HIV infection);
4. The presence of any active, known or suspected autoimmune disease (such as, but not limited to, interstitial pneumonia, uveitis, enteritis, hepatitis, arthritis, nephritis, hypophysitis, hyperthyroidism, hypothyroidism, etc.); Medical history of vitiligo; asthma which requires bronchodilators for medical intervention;
5. Active infection requiring systemic treatment;
6. Previously treatment with PD-1 and/or PD-L1, or CTLA-4 antibody, or other medications targeting immunomodulatory receptors;
7. Patients with grade>2 unrelieved toxic reactions (based on National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0) caused by any previous treatment;
8. With a history of myocardial infarction,stroke, unstable angina, decompensated heart failure, or deep vein thrombosis;
9. Long-term uncured wounds or fractures; Major surgery or severe traumatic injury, fracture or ulcer within 4 weeks;
10. Pregnant or lactating women;
11. With metastatic diseases;
12. Liver/renal insufficiency;
13. Those who have a history of psychotropic drug abuse and cannot get rid of it or those with mental disorders;
14. Those who have participated in clinical trials with other drugs within 4 weeks;
15. Patients with concomitant diseases or abnormal test results which interfere with the ability to receive anticancer therapy judged by the investigator;
16. Patients could not gain the maximum benefit from this study judged by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year progress free survival rate | up to 3 years
  Progression-free survival (PFS) is defined as the time between entry into the study and progression of the tumor (in any respect) or death (from any cause).
side effect rate | up to 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective response rate(ORR) | 3 months, after chemoradiotherapy
  ORR is defined as the proportion of patients with CR or PR, assessed by RECIST v1.1 per independent central radiologic review.
3-year overall survival rate | up to 3 years
  overall survival rate（OS）is calculated from the date of entry into the study to the date of death or the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: fang wu, M.D., Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No